CLINICAL TRIAL: NCT07144774
Title: The Effectiveness of Wearable Devices on Health Promotion in Individuals With Diabetes Mellitus
Brief Title: Wearable Devices on Health Promotion in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific University (Other)
Responsible Party: Principal Investigator, Eliza Wu, Assistant Professor, Pacific University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2032697-1 / 048-23
Record Dates: First submitted 2025-08-13; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Diabetes (DM)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group were provided with a Fitbit wrist-worn device (Inspire 2® activity tracker) at baseline.
  Interventions: Device: Fitbit wrist-worn Inspire 2® activity tracker (Fitbit Inc., San Francisco, CA, USA)
- Control group (No Intervention): Participants in the control group did not receive a wearable device but were instructed to carry their smartphones throughout the day to enable step tracking via the MobileTrack feature.

INTERVENTIONS:
Device: Fitbit wrist-worn Inspire 2® activity tracker (Fitbit Inc., San Francisco, CA, USA) — Visual feedback of the physical activity level
  Arms: Intervention group

SUMMARY:
This proposed study involves human participants who will be prospectively randomized into either 1) intervention group with a activity tracker or 2) control group without an activity tracker. In addition, the proposed study is designed to evaluate the effect of using an activity tracker on cardiovascular health in the study participants.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. diagnosed with type 2 diabetes (HbA1c ≥ 6.5% or fasting plasma glucose ≥ 126 mg/dL)
3. willing to link a fitness tracker (Fitbit®) App to their own smartphone

Exclusion Criteria:

1. are unable to walk without assistive devices,
2. are current smokers,
3. are pregnant or breastfeeding,
4. already engage in ≥ 150 minutes of moderate-to-vigorous physical activity per week,
5. have any medical conditions (e.g., musculoskeletal diseases, cognitive dysfunction) that will interfere with physical activity,
6. undergo any insulin treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Step Counts | 4 weeks
  Daily step counts (steps/day) were collected using the activity tracker and mobile app.
Walking distance | 4 weeks
  Daily walking distance (meters/day) was collected using the activity tracker and mobile app.
Energy expenditure | 4 weeks
  Daily energy expenditure (calories/day) was collected using the activity tracker and mobile app.
Time spent in physical activity and sedentary behaviors | 4 weeks
  Time (hours : minutes) spent in physical activity and sedentary behaviors in a week was collected using the Global Physical Activity Questionnaire (GPAQ). The GPAQ consists of 16 questions designed to estimate an individual's level of physical activity in 3 domains (work, transport, and recreational activities) and time spent in sedentary behavior.
Blood pressure | 4 weeks
  Brachial systolic and diastolic blood pressure (mmHg) was collected using an automated sphygmomanometer. Pulse pressure and mean arterial pressure were calculated from systolic and diastolic blood pressure.
Augmentation index | 4 weeks
  Augmentation index (%), as an indicator of arterial stiffness, was assessed using applanation tonometry (SphygmoCor®, AtCor Medical, Sydney, Australia).
Pulse wave velocity | 4 weeks
  Pulse wave velocity (meter/second), as an arterial stiffness indicator, was assessed using applanation tonometry (SphygmoCor®, AtCor Medical, Sydney, Australia).
Subendocardial viability ratio | 4 weeks
  The subendocardial viability ratio (SEVR) was measured as an index of myocardial perfusion and coronary supply-demand balance, using applanation tonometry (SphygmoCor®, AtCor Medical, Sydney, Australia).

SECONDARY OUTCOMES:
Metabolic measures | 4 weeks
  Fasting glucose level
Body mass index | 4 weeks
  Body weight (kilograms) and height (meters) were measured and used to calculate body mass index (kg/m^2).
Waist-to-hip ratio | 4 weeks
  Waist and hip circumferences (centimeters) were measured and used to calculate the waist-to-hip ratio.

OTHER OUTCOMES:
Quality of life via survey | 4 weeks
  The quality of life was assessed using the 36-Item Short Form Health Survey (SF-36). The SF-36 consists of eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
  All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Pei Tzu Wu, Principal Investigator — Pacific University
Locations (1):
- Pacific University, Hillsboro, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and statistical analysis plan will be shared.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Azar KM, Koliwad S, Poon T, Xiao L, Lv N, Griggs R, Ma J. The Electronic CardioMetabolic Program (eCMP) for Patients With Cardiometabolic Risk: A Randomized Controlled Trial. J Med Internet Res. 2016 May 27;18(5):e134. doi: 10.2196/jmir.5143. PMID 27234480
- [Background] Lystrup R, Carlsen D, Sharon DJ, Crawford P. Wearable and interactive technology to share fitness goals results in weight loss but not improved diabetes outcomes. Obes Res Clin Pract. 2020 Sep-Oct;14(5):443-448. doi: 10.1016/j.orcp.2020.08.006. Epub 2020 Sep 3. PMID 32891527
- [Background] Hodkinson A, Kontopantelis E, Adeniji C, van Marwijk H, McMillian B, Bower P, Panagioti M. Interventions Using Wearable Physical Activity Trackers Among Adults With Cardiometabolic Conditions: A Systematic Review and Meta-analysis. JAMA Netw Open. 2021 Jul 1;4(7):e2116382. doi: 10.1001/jamanetworkopen.2021.16382. PMID 34283229

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Wearable Device on Health Promotion in Diabetes (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT07144774/Prot_SAP_000.pdf